CLINICAL TRIAL: NCT05781555
Title: A Prospective, Open Label, One Arm Study for a Compassionate Use of Diffusing Alpha Radiation Therapy
Brief Title: A Study of Diffusing Alpha Radiation Therapy for Target Treatments of Malignant Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP- ALL-00
Record Dates: First submitted 2023-02-26; First posted 2023-03-23 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-05

CONDITIONS: Malignant Tumor
Keywords: Tumor; Malignant Tumor; Cancer; Brachytherapy; Alpha emitting radiation; Compassionate treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: Experimental: DaRT seeds

INTERVENTIONS:
Device: Experimental: DaRT seeds — DaRT source will be inserted using preplanned radiotherapy parameters and reassessed by volumetric imaging 2-3 weeks after placement and then removed. The study objectives are to collect data on the general safety and efficacy of DaRT among patients who do not fit the entry criteria of existing investigational trials.

SUMMARY:
This study is a Compassionate clinical study for the treatment of Malignant Tumors. The primary endpoint of the study is to assess the frequency, severity and causality of acute adverse events related to the DaRT treatment. Adverse events will be assessed and graded according to Common Terminology and Criteria for Adverse Events (CTCAE) version 5.0. The secondary endpoint is to assess the tumor response to DaRT treatment assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1) 3 months after DaRT seed insertion.

DETAILED DESCRIPTION:
This is an Open label, one arm, prospective study for Compassionate use for the treatment of malignant tumors. The study objectives are to collect data on the safety and efficacy of DaRT among patients who do not fit the entry of existing investigational trials.

The primary endpoint of the study is to assess the frequency, severity and causality of acute adverse events related to the DaRT treatment. Adverse events will be assessed and graded according to Common Terminology and Criteria for Adverse Events (CTCAE) version 5.0. The secondary endpoint is to assess the tumor response to DaRT treatment assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1) 3 months after DaRT seed insertion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with any malignancy
* Subjects with a tumor size ≤ 7 centimeters in the longest diameter
* Subjects over 18 years old
* Subjects' life expectancy is more than 6 months
* Women of childbearing potential (WOCBP) will have evidence of negative pregnancy test and are required to use an acceptable contraceptive method to prevent pregnancy for 3 months after treatment.
* Subjects/Surrogate decision maker are willing to sign an informed consent form

Exclusion Criteria:

* Known hypersensitivity to any of the components of the treatment.
* Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 12 months.
* Any medical or psychiatric illness which in the opinion of the investigator would compromise the patient's ability to tolerate this treatment or interfere with the study endpoints.
* Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT.
* Patients must agree to use adequate contraception (vasectomy or barrier method of birth control) prior to study entry, for the duration of study participation and for 3 months after discontinuing therapy.
* High probability of protocol non-compliance (in opinion of investigator).
* Subjects/Surrogate decision maker not willing to sign an informed consent.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
To assess the frequency, severity and causality of acute adverse events. | From Day 0 (DaRT insertion )
  The primary endpoint of the study is to assess the frequency, severity and causality of acute adverse events related to the DaRT treatment. Adverse events will be assessed and graded according to Common Terminology and Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
To assess the tumor response to DaRT treatment | 3 months after DaRT seed insertion
  The secondary endpoint is to assess the tumor response to DaRT treatment assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Aron Popovzer, MD, Principal Investigator — Hadassah University Hospital - Ein Kerem
Locations (1):
- Hadassah Ein Kerem, Jerusalem, Israel